CLINICAL TRIAL: NCT06731569
Title: Evaluation of the Lateral Window Approach of Maxillary Sinus Floor Augmentation Using a Newly Designed Advanced Intelligence Drill: a Randomized Clinical Trial
Brief Title: Advanced Intelligence Driven Drill for Maxillary Sinus Augmentation in Patients with Severe Bone Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-H-0126-D-M-0560
Record Dates: First submitted 2024-11-26; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-12

CONDITIONS: Maxillary Sinus Floor Augmentation
Keywords: dental implant; Advanced intelligence drill; osteotomy; maxillary sinus floor augmentation; schneiderian membrane; perforation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups, and each group receives a specific intervention:
  Group A: Traditional rotary drill. Group B: AI drill.
  Each group is treated independently, and the outcomes are compared at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Traditional rotary drill (Control Group) (Active Comparator): Participants in this arm will undergo Maxillary Sinus Floor Augmentation (MSFA) using the traditional rotary drill. The procedure involves preparing the lateral window with a rose-head bur, ensuring precision and irrigation to minimize trauma. The traditional drill is widely used in clinical practice but requires significant skill to avoid complications like Schneiderian membrane perforation.
  Interventions: Device: Traditional rotary instrument
- AI-powered drill (Intervention Group) (Experimental): Participants in this arm will undergo MSFA using a newly designed AI-powered drill. This innovative drill automatically stops rotation upon detecting the Schneiderian membrane, reducing the risk of perforation. The intervention also includes the use of specialized hydraulic pressure to aid in membrane elevation and preparation of the lateral window for grafting. The AI drill aims to enhance precision, efficiency, and safety during the procedure.
  Interventions: Device: Advanced intelligence drill

INTERVENTIONS:
Device: Advanced intelligence drill — The AI drill is an innovative surgical tool designed specifically for Maxillary Sinus Floor Augmentation (MSFA) procedures. It incorporates advanced technology to enhance safety, precision, and efficiency during lateral window preparation.
  It has an Automated Pressure-Sensing Mechanism which makes the drill automatically stops rotating when it detects contact with the Schneiderian membrane, minimizing the risk of perforation.
  The OLA kit consists of Hydraulic Lift which is compatibility with the drill connected to a saline-filled syringe to gently elevate the Schneiderian membrane from the sinus floor.
  It involves a Multi-Step Drilling Process using different drill tips designed each for a specific task including the pilot drill for initial window creation and the non-cutting ball-end drill for lateral wall thinning and smoothing.
  It works at a controlled high-Speed Performance of 6000 RPM with irrigation system included.
  Other Names: OLA Kit
  Arms: AI-powered drill (Intervention Group)
Device: Traditional rotary instrument — Traditional Rotary Drill
  The traditional rotary drill is a commonly used surgical tool in Maxillary Sinus Floor Augmentation (MSFA) procedures, employing conventional drilling techniques for lateral window preparation. It is a widely recognized method due to its accessibility and effectiveness in skilled hands.
  It Uses a rose-head bur attached to a surgical straight handpiece that operates at speeds of 800-1200 RPM with irrigation to prevent overheating and ensure efficient bone cutting.
  It is a manual operator control that requires the surgeon's skill and experience to control the depth and force of drilling. And relies on visual and tactile feedback to identify when the Schneiderian membrane is close to exposure.
  It is versatile and can be adapted to varying bone densities and anatomical complexities. It is effective for creating the window for sinus access.
  It comes with an irrigation system to avoid necrosis of the bone.
  Other Names: Rosehead Bur
  Arms: Traditional rotary drill (Control Group)

SUMMARY:
Study Summary

The goal of this clinical trial is to evaluate whether a newly designed Advanced Intelligent drill can improve the safety and effectiveness of Maxillary Sinus Floor Augmentation (MSFA) procedures in adults with insufficient bone height in the posterior maxilla for dental implants.

The main questions it aims to answer are:

* Can the AI drill reduce the risk of Schneiderian membrane perforation compared to traditional drilling methods?
* Does the AI drill improve the efficiency of window preparation during the procedure?

The researcher compares the outcomes of participants treated with the AI drill to those treated with a traditional rotary drill to see if the AI drill leads to fewer complications (less membrane perforations, bleeding and postoperative complications) and better surgical outcomes.

Participants will:

* Undergo MSFA using either the AI-powered drill or the traditional rotary drill.
* Attend follow-up appointments to monitor healing and outcomes, including imaging and clinical evaluations.

This study hopes to advance surgical techniques for safer and more effective preparation for dental implants.

DETAILED DESCRIPTION:
This study investigates a new technology designed to make dental procedures safer and more effective. Specifically, it focuses on a the lateral approach of Maxillary Sinus Floor Augmentation (MSFA), used to prepare the insufficient maxilla for dental implants in areas with low bone height. The study compares a traditional drilling method to an advanced intelligence drill to determine which is better at reducing complications and improving outcomes.

{Purpose of the Study}

The goal is to evaluate if the advanced intelligent drill can:

* Reduce the risk of Schneiderian membrane perforation
* Make the procedure (bony window opening) quicker and easier for both patients and dentists.
* Provide better conditions for bone graft site and for dental implants.

{Participants}

In the study, all participants presented with less than 5 mm of bone height in the posterior maxilla and in need of MSFA procedure using the lateral window approach.

All participants are healthy patients without major systemic diseases (like uncontrolled diabetes or recent cancer treatments) who need dental implants but have insufficient bone height in the upper jaw.

Participants with the following were excluded from the study:

* Active sinus infections.
* Large cysts or tumors in the jaw.
* Recently had sinus surgeries.

{Study Methods}

Participants were split into two groups:

Group A: Traditional Drilling Group: Used a standard dental drill to prepare the bony window.

Group B: AI Drill Group: Used the new AI-powered drill that stops automatically when it touches the schneiderian membrane, reducing the chance of damage.

All procedures were done under local anesthesia, and patients were monitored closely before, during, and after surgery.

Clinical and Radiographic diagnosis of the cases were done following a precise protocol by the operator.

Pre-operative diagnosis and planning of all cases is fundamental to avoid intra- and post- operative complications. Many factors are to be evaluated during this time. A MSFA checklist is put in place.

All the procedures are achieved with the full knowledge and consent of the patient. A written informed consent is obtained for each patient included in this study.

{Surgery}

PRE-SURGICAL PHASE

Investigations and Primary Evaluation

1. A proper diagnosis and subsequent proper case selection must be achieved. A clinical and radiographic treatment planning using a Cone Beam Computer Tomography (CBCT) is mandatory. This diagnostic tool is essential in this region to provide precision in the measurement of the residual bone height and its density. It also adds information about the anatomy of the maxillary sinus, the presence of any pathologies and the presence of a septa.
2. The residual bone level is measured from the CBCT: from the most inferior border of the maxillary sinus to the alveolar crest in a sagittal direction.
3. The Schneiderian membrane thickness is measured from the CBCT.

SURGICAL PHASE

The surgery is performed by the same surgeon. Precautions are taken to operate in sterile conditions. All procedures are performed under local anesthesia (articaine 4% in combination with epinephrine).

Procedure:

* Raise a full thickness mucoperiosteal flap with vertical incision exposing the alveolar ridge and the lateral wall of the maxillary sinus
* Perform the lateral window osteotomy using a rose-head bur or A.I drill. In the procedure using the OLA kit: the osteotomy is initiated using the A.I drill followed by the aqua lifter connected to a disposable syringe which is indicated to infuse physiological saline of 1.0-1.5 cc to preliminarily lift the Schneiderian membrane.
* Carefully elevate the sinus membrane using the special hand instruments
* Carry the Valsalva maneuver to make sure the sinus membrane is fully elevated and has no perforations
* The sinus floor is augmented using xenograft through the lateral window to fill the sub antral space created then covered with a resorbable collagen membrane.
* The wound is sutured by 4/0 PGA sutures

POST-OPERATIVE CARE

* Antibiotic therapy (amoxicillin + clavulonic acid 1000 mg BID) is prescribed for the next 7 days along with Non-Steroidal Anti-Inflammatory Drug (NSAID) (Ibuprofen 400 mg BID) for 5 days for pain and swelling.
* The patient is advised not to brush the area or apply pressure by eating on it. He is also advised to avoid smoking, blowing their noise and other activities that may increase the sinus pressure for one week post operative.
* Sutures are removed 7 to 10 days after surgery.

FOLLOW UP

The maxillary implants are not to be placed until a 6-months healing time has elapsed. Thus, a follow up is done at 1 months, 3 months and 6 months after MSFA procedure. The bone level assessed and measured via CBCT imaging at 6 months post-operative.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are free from any systemic disorders
2. Residual bone height ≤ 5 mm
3. Absence of any infections in the maxillary sinus to be treated.
4. Highly co-operative and motivated patients who follow the pre- and post- operative care instructions.
5. Adequate vertical space indicated for implant placement and subsequent prosthesis (minimum of 4-5 mm)

Exclusion Criteria:

1. Participants with uncontrolled systemic conditions including Diabetes, Hypertension and Hyperthyroidism
2. Participants currently undergoing chemotherapy or radiotherapy.
3. Participants on current bisphosphonate therapy or on medication that could interfere with the sinus lift procedure.
4. Presence of sinus infection
5. Presence of a neoplasm or a large cyst of the sinus
6. Participants who previously underwent a Caldwell-Luc surgery for the same Study Interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Duration of the procedure | From the beginning of anaesthesia injection until the last suture is done
  Duration of the procedure a stopwatch in minutes and seconds will be used to time in minutes and seconds the procedure from the beginning of anaesthesia injection until the last suture is done.
Duration of Osteotomy/Window preparation | from the moment the drilling starts the osteotomy preparation till the complete window is formed
  A stopwatch will be used to time in minutes and seconds from the moment the drilling starts the osteotomy preparation till the complete window is formed.
Clinical Schneiderian membrane thickness | immediately after osteotomy is done
  During surgery: clinically by the surgeon's visual assessment according to the membrane translucency (Clear Translucent or Thick) by Score 0 and 1
Radiographic Schneiderian membrane thickness | Pre-operative
  Pre-operatively assessed by radiographic imaging (CBCT) in millimeters
Perforation of the Schneiderian membrane | During the surgery immediately when perforation occurs
  Perforation of the Schneiderian membrane: It is measured by a periodontal probe in millimeters

SECONDARY OUTCOMES:
Excessive Bleeding | During the surgery when bleeding occurs
  Assessed during the procedure (presence/abscence score)
Manipulation of the Drill used | From the beginning of the drilling until end of drilling
  assess its ease of access intra-operatively (Easy: 1, Hard: 0)
Satisfaction of Drill to operator | from the beginning of the drilling until the end of the drilling
  Subjective assessment by giving a score 0 for not satisfied and 1 for satisfied
Baseline Residual Bone Height | Pre-operative
  Measured from CBCT in millimeters: from the most inferior border of the maxillary sinus to the alveolar crest in a sagittal direction
Post-operative Bone Volume Gain | immediately after surgery and at 6 months post-operative
  Measured on the CBCT immediately after surgery in millimeters and again 6 months post-operative at the follow up
Post-operative Water Height (WH) in the sinus | Immediately after surgery
  Measure in millimeters on the CBCT immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nayer Aboelsaad, Professor, Study Chair — Beirut Arab University
Locations (1):
- Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
The following individual participant data will be shared for this clinical study:
  1. Pre-Operative Assessments:
     * Cone Beam Computed Tomography (CBCT) measurements of residual bone height and Schneiderian membrane thickness.
     * Presence or absence of anatomical variations (e.g., bony septa, posterior superior alveolar artery).
  2. Intraoperative Data:
     * Duration of procedure and window preparation time.
     * Incidence of Schneiderian membrane perforation.
     * Details of bleeding events (if any), including management approaches.
  3. Postoperative Outcomes:
     * Graft volume and resorption rates.
     * Bone gain at the surgical site (immediate and at 6 months follow-up).
Supporting Information: SAP, CSR